CLINICAL TRIAL: NCT04915404
Title: A Multicenter, Open-Label Study of the Efficacy, Safety, and Pharmacokinetics of Intravenously Infused Berubicin in Adult Patients With Recurrent Glioblastoma Multiforme (WHO Grade IV) After Failure of Standard First Line Therapy
Brief Title: Berubicin in Adult Patients With Recurrent Glioblastoma Multiforme (WHO Grade IV)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: WPD Pharmaceuticals Sp. z o.o. (Industry)
Collaborators: Worldwide Clinical Trials (Other); National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WPD-201
Record Dates: First submitted 2021-02-23; First posted 2021-06-07 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Recurrent Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pK Assessment of Berubicin and its active metabolite (Experimental): The first 18 patients will undergo a pK assessment of Berubicin and it's active metabolite Berubicinol during the dosing days of the first two cycles. After 18 patients are done n intern analysis will new performed.
  Interventions: Drug: Berubicin Hydrochloride

INTERVENTIONS:
Drug: Berubicin Hydrochloride — Berubicin intravenously infused will be administered at a dose of 7.1 mg/m2 as free base (equivalent to 7.5 mg/m2 Berubicin HCl) as a 2-hour intravenous (IV) infusion once daily for 3 consecutive days followed by 18 days off study drug (each cycle = 21 days).

SUMMARY:
This is a multicenter, open-label, Phase 1b/2 efficacy and safety study of Berubicin utilizing a Simon's 2-stage design to confirm the efficacy (or futility) of a single arm of Berubicin treatment, administered at the recommended Phase 2 dose (RP2D) identified in Phase 1 studies (7.5 mg/m2 Berubicin HCl), on the endpoint of ORR in up to approximately 61 patients. A central reader will determine the radiologic responses for each patient according to m RANO criteria. The responder criteria for this Simon's design will be based on objective response criteria defined as individual patients achieving CR or PR per m-RANO criteria within 6 months from baseline.

DETAILED DESCRIPTION:
The planned minimum duration of the study for an individual patient is approximately 11 weeks as follows:

* A 4-week Screening Period
* A 3-week Treatment Period (ie, one 3 week treatment cycle)
* A 4-week End-of-Treatment follow-up Period after the last dose The 3-week treatment cycles may be repeated in the absence of clinical and/or neurological deterioration, or unacceptable toxicity, and as long as both the patient and investigator agree that further therapy is in the patient's best interest.

After the End-of-Treatment follow-up visit, patients will enter a Post-Study follow-Up Period of up to approximately 2 years.

ELIGIBILITY:
Patients will be eligible for the study if they meet all of the following inclusion criteria and none of the exclusion criteria.

Inclusion criteria

1. Written informed consent prior to any study-related procedure, and willing and able to comply with the protocol and aware of the investigational nature of this study.
2. At least 18 years of age.
3. A diagnosis of GBM (WHO Grade IV) confirmed by:

   1. Archived paraffin-embedded tissue (approximately 10 unstained slides or a tumor block) from initial resection for local review of tumor diagnosis OR
   2. A tumor tissue form indicating diagnosis from initial resection of glioblastoma completed and signed by a pathologist and/OR
   3. Tumor tissue from re-resection, managed as above (a OR b)
4. Measurable disease is required with documented unequivocal evidence of tumor recurrence or progression following prior therapy, confirmed by the following:

   1. Recurrent GBM as documented by the principal investigator (PI). In case of recent interim debulking surgery, the histopathological verification of the resected tissue as recurrent tumor automatically qualifies the patient as eligible for the trial.
   2. KPS reduction of 10 units while on stable or increasing doses of corticosteroids as documented by the PI
   3. Subject MRI meets at least two of the following three criteria as determined by central review:

      1. Presence of measurable disease: the lesion is ≥10 mm in both maximum perpendicular diameters
      2. Evidence of unequivocal tumor recurrence or progression following prior therapy as determined by a 10% increase in the sum of the products of perpendicular diameters of the contrast-enhancing lesions
      3. Substantial increase in the perilesional oedema as shown in T2/FLAIR images.
5. All contrast enhancing disease is located supratentorially
6. O[6] methylguanine-DNA methyltransferase (MGMT) methylation status must be available, or able to be determined from existing tumor tissue; results of routinely used methods for MGMT methylation testing (e.g., methylation-specific polymerase chain reaction [MSPCR] or quantitative polymerase chain reaction [PCR]) are acceptable.
7. No more than 1 prior line of treatment (e.g., surgery followed by radiation with concomitant chemotherapy, followed by adjuvant chemotherapy is considered as 1 line of treatment). A second debulking surgery during the first line treatment is acceptable.
8. Recovery from toxicity/side effects of all prior therapy to Grade 1 or less, subject to the investigator's discretion, except for alopecia; the following time intervals from previous treatments are required to be eligible:

   1. 12 weeks from the completion of radiation (to reduce risk of pseudoprogression), unless progression is confirmed by biopsy
   2. 4 weeks from the end of any previous chemotherapy or 6 weeks after the end of treatment with nitrosoureas
   3. 4 weeks from any major surgery (maximal debulking surgery, either gross total resection or partial resection) or significant traumatic injury, and any surgery incisions or wounds must be completely healed
9. A stable or decreasing dose of corticosteroids (or none) for brain edema for at least 5 days prior to baseline MRI and enrollment in the study as confirmed by the PI.
10. Immunosuppressive therapies allowed include the use of topical, inhalational, ophthalmic, or intra-articular glucocorticoids, or the use of physiologic replacement doses of glucocorticoids.
11. Eligible for chemotherapy based on adequate bone marrow function and organ function within 2 weeks of study treatment as defined by the following laboratory guidelines, subject to the investigator's discretion:

    1. Hematopoietic function: total white blood cell (WBC) count ≥3000/mm³, absolute neutrophil count (ANC) ≥1500/mm³, platelet count ≥75,000/mm³, hemoglobin ≥10 g/dL
    2. Hepatic function: bilirubin ≤1.5 × the upper limit of normal (ULN) (excluding Gilberts Syndrome, for which bilirubin must be ≤4 × ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 × ULN, and alkaline phosphatase ≤2.5 × ULN
    3. Renal function: serum creatinine ≤1.5 × ULN or for patients with creatinine levels above the ULN, or estimated creatinine clearance of ≥60 mL/min/1.73 m2, calculated using the Cockcroft Gault formula
    4. Activated partial thromboplastin time (aPTT) ≤1.5 × ULN.
12. Women of childbearing potential must agree to practice a highly effective method of contraception beginning at least 28 days before the start of treatment until at least 6 months after the last dose of study drug. Male study patients and their female sexual partners of childbearing potential must agree to practice a highly effective method of contraception starting from the time of informed consent until at least 3,5 months (no less than 104 days) after the last dose of study drug.

    1. A woman of childbearing potential is defined as a woman who is not permanently sterilized or postmenopausal. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.
    2. Women of childbearing potential must have a negative serum or urine pregnancy test.
    3. A highly effective method of birth control is defined as one which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. For patients using a hormonal contraceptive method, information regarding all medications being administered to the patient and their potential effect on the contraceptive should be addressed.
13. Patients with prior malignancies must be disease-free for ≥5 years. However, curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; or prostate cancer curatively treated at the time of screening is allowed.

Exclusion Criteria

1. Unable or not willing to comply with the protocol regulations.
2. Any additional concurrent radiation therapy or chemotherapy (including but not limited to temozolomide [TMZ]) for recurrent or progressive GBM after a first line treatment.
3. Prior treatment with bevacizumab.
4. The presence of IDH mutation prior to enrollment
5. Screening MRI showing a mass effect defined as significant compression of the ventricular system and/or a midline shift (≥10 mm) as determined by central MRI review.
6. Any condition (medical, social, psychological) that would prevent adequate information and follow-up, including but not limited to clinically relevant psychiatric disorders, legal incapacity, dementia, or altered mental status.
7. Presence of poorly controlled seizures, defined as occurring despite standard of care (SOC) or requiring hospitalization.
8. Widespread or focal leptomeningeal disease measuring ≥10mm by ≥10mm.
9. Prior anthracycline cumulative dose more than 550 mg/m2.
10. Heart disease:

    1. LVEF <50%
    2. Unstable angina
    3. Congestive heart failure with New York Heart Association (NYHA) classification of 3 or 4
    4. Patients with baseline QT/QTc interval >480 msec, a history of additional risk factors for torsades de pointes (TdP) (e.g., heart failure, hypokalemia, family history of long QT syndrome) and using concomitant medications that significantly prolong the QT/QTc interval
    5. History of myocardial infarction within 12 months of enrollment.
11. Uncontrolled hypertension (systolic blood pressure [BP] >150 mmHg and/or diastolic BP >100 mmHg).
12. Known to be positive for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV), human immunodeficiency virus (HIV), coronavirus disease-2019 (COVID-19) or any other acute viral, bacterial, or fungal infection (testing not required unless symptomatic or suspected disease).
13. Any other uncontrolled intercurrent medical conditions, including but not limited to diabetes mellitus or chronic obstructive pulmonary disease that have not been well controlled by medical management over the prior 3 months are ineligible unless approved by the sponsor.

WPD reserves the right to deny any patient enrollment based upon any potential safety concern(s) or factors that could confound the study results.

Note: Investigator (PI or designee) review of all screening assessment results is required to determine eligibility prior to Berubicin administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) | 6 months
  To confirm the efficacy (or futility) of Berubicin treatment on objective response rate (ORR) defined as CR or PR per modified Response Assessment in Neuro-Oncology (m RANO) criteria in patients with GBM (World Health Organization [WHO] Grade IV) that has recurred after standard initial therapy, based on Simon's 2-stage design

SECONDARY OUTCOMES:
• To confirm the safety profile of Berubicin that was characterized during Phase 1 studies and assess the effect of Berubicin on event-free survival (EFS) | 6 months
  • To assess the effect of Berubicin on event-free survival (EFS) defined as the length of time from the initiation of study drug administration to stable disease , disease progression, death, or discontinuation of treatment for any reason (eg, toxicity, intolerance, disease-related conditions, or failure to respond). Safety will be monitored by a safety review committee (SRC). The SRC will review PK and safety data from the first 2 cycles of treatment for the first approximately 18 patients (i.e., Stage 1) of this study
• To confirm the pharmacokinetic (PK) profile of Berubicin and its metabolite, berubicinol, that was characterized during Phase 1 studies | 6 months
  intensive pK assessment of Berubicin and it's active metabolite will be performed during the dosing days of the first two cycles , this will be folowed by an interim analysis at 18 patients time point.Plasma samples will be collected from the first approximately 18 patients enrolled, and concentrations of Berubicin and its metabolite, berubicinol, will be measured
• To assess the effect of Berubicin on disease control rate (DCR) defined as CR or PR or stable disease [SD] per m-RANO criteria in patients with GBM after failure of standard first line therapy | 12 months
  Screening/baseline MRI scans will be evaluated by a central reader for validation of eligibility and documentation of initial measurements. During the Treatment Period, the baseline scan will be compared with scans at 6-week (2-cycle) intervals for evaluation of disease by the investigator as well as the central reader according to m-RANO criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne Klinika Onkoligii i Radioterapii, Gdansk
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie,Państwowy Instytut Badawczy w Warszawie,Klinika Nowotworów Głowy i Szyi, Warsaw

IPD SHARING:
Plan to Share IPD: No